CLINICAL TRIAL: NCT04997720
Title: ANALYSIS OF THE IMPACT ON THE MICRO SURGICAL TECHNIQUE IN RESIDENTS AFTER A THEORETICAL-PRACTICAL COURSE OF MICROSURGERY: A SINGLE GROUP STUDY
Brief Title: Impact of the Microsurgical Technique After a Theoretical-practical Course in Microsurgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas José de San Martín (Other)
Responsible Party: Principal Investigator, Marcos Ezequiel Yasuda, Medical Doctor, Hospital de Clinicas José de San Martín
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1092-21
Record Dates: First submitted 2021-07-03; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Medical Training; Microsurgery; Education
Keywords: Academic training; Capacity evaluation; Continuing medical education; Neurosurgery

STUDY DESIGN:
Masking Description: The evaluation will be in charge of the teacher who will record the practical evaluation. Then all the videos will be analyzed blindly by a neurosurgeon with experience in microsurgery. Statistical analyzes will also be analyzed blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Other): The course will be theoretical-practical, lasting eight hours, divided into two meetings with a theoretical class and practical exercises in microsurgery of increasing complexity. The course will also have an initial and final evaluation.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — Each course will consist of:
  1. Initial evaluation
  2. Theoretical tutorial
  3. Training with exercises of increasing complexity.
  4. Final evaluation.

SUMMARY:
A single group study will be carried out in the Microsurgery Laboratory, Neurosurgery Department, Hospital de Clínicas, and the Center for Microsurgical Skills of the Argentine Association of Neurosurgery. The objective of the study is to evaluate the effect of theoretical-practical course learning in neurosurgery and plastic surgery residents.

DETAILED DESCRIPTION:
Introduction: In the second half of the 20th century, the use of the surgical microscope became popular in neurosurgery. In the last twenty years, simulation has gained worldwide acceptance as a teaching tool in medicine, especially microsurgery. For this, various training models have been created.

Objective: To evaluate the effect of the theoretical-practical course learning in neurosurgery and plastic surgery residents.

Materials and methods: A single group study will be carried out in the Microsurgery Laboratory, Neurosurgery Department, Hospital de Clínicas, and the Center for Microsurgical Skills of the Argentine Association of Neurosurgery. Medical doctors of both genders will be included in the first three years of neurosurgical or plastic surgery training from any center in Argentina. The course will be theoretical-practical, lasting eight hours, divided into two meetings with a theoretical class and practical microsurgery exercises. It will be supervised by teachers microsurgery experienced. An Initial and final evaluation will be carried out and the scores obtained between both theoretical and practical evaluations will be compared. In the practical evaluations, the time and the SMART scale will be analyzed. Categorical variables will be reported as absolute and relative numbers. The normality of the data will be verified by the Kolmogorov-Smirnov test. Continuous variables will be reported as mean and standard deviations or median and interquartile ranges. Student's t test, Mann-Whitney U test will be used to compare means, when appropriate, according to the distribution of variables. The categorical variables will be compared with the χ2 test.

ELIGIBILITY:
Inclusion Criteria:

* Doctors in the first three years of neurosurgical training or plastic surgery in any center in Argentina.
* Both gender will be included without age limit.

Exclusion Criteria:

* Participants who do not complete the entire course will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Change of Quality of the execution of the suture | Change from baseline of Score Stanford Microsurgery and Resident Training Scale (SMART)through study completion, an average of 8 hours of training
  The process of executing the suture will be evaluated using the Stanford Microsurgery and Resident Training Scale (SMART) (9 to 45, higher scores mean a better outcome)
Change of Time of the execution of the suture | Change from baseline through study completion, an average of 8 hours of training
  The time in seconds required to complete the evaluation
Change of Theoretical knowledge | Change from baseline through study completion, an average of 8 hours of training
  A theoretical evaluation of ten multiple-choice questions

SECONDARY OUTCOMES:
The correlation between the year of residence and the changes in the results of the theoretical evaluation of ten multiple-choice questions. | Change from baseline after 8 hours of training
  To identify if the year of residence influences the theoretical evaluation of ten multiple-choice questions.
The correlation between the year of residence and the changes in the results of the time in seconds required to complete the evaluation. | Change from baseline after 8 hours of training
  To identify if the year of residence influences the time in seconds required to complete the evaluation
The correlation between the year of residence and the changes in the process of executing the suture will be evaluated using the Stanford Microsurgery and Resident Training Scale (SMART) (9 to 45, higher scores mean a better outcome) | Change from baseline after 8 hours of training
  To identify if the year of residence influences the process of executing the suture will be evaluated using the Stanford Microsurgery and Resident Training Scale (SMART) (9 to 45, higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Ezequiel Yasuda, Caba, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No